CLINICAL TRIAL: NCT00485472
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Trial to Assess the Efficacy and Safety of 400mg/Day Lacosamide in Subjects With Osteoarthritis of the Knee
Brief Title: Trial to Assess Efficacy and Safety of Lacosamide in Subjects With Osteoarthritis of the Knee
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Based on the outcome of the planned first interim analysis, it was decided not to continue the trial. No safety concerns were identified.
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SP0905; 2006-005048-97 (EudraCT Number)
Record Dates: First submitted 2007-06-12; First posted 2007-06-13 (Estimated); Results first posted 2009-09-22 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-07

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; lacosamide; VIMPAT
MeSH Terms: conditions — Osteoarthritis | interventions — Lacosamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lacosamide (Experimental): lacosamide (LCM)
  Interventions: Drug: lacosamide
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: lacosamide — 50 or 100mg tablet, 400mg daily, for 12 weeks
  Other Names: VIMPAT
  Arms: Lacosamide
Other: Placebo — 50 or 100mg tablet, 400mg daily, for 12 weeks, matched to Lacosamide
  Arms: Placebo

SUMMARY:
The purpose of this trial is to evaluate the effectiveness, safety and tolerability of lacosamide (LCM) 400mg/day in treating the signs and symptoms of osteoarthritis of the knee.

DETAILED DESCRIPTION:
LCM is an investigational drug that is being studied as a treatment in male and female patients who are diagnosed with osteoarthritis of the knee and require therapeutic doses of NSAIDs, COX-2 NSAIDs and/or paracetamol. This trial will be conducted exclusively in Europe.

The study has an adaptive 3-stage group sequential design.

The trial will last a total of 17 weeks. There will be a 2 week period to wean off current medication, followed by a 4 week period where the patient will receive placebo (inactive drug) or gradually increasing doses of LCM up to the target dose of 400mg/day. The target dose or placebo will be maintained for 8 weeks followed by a 1 week reduction period then a 2 week safety follow up period.

The last subject is expected to be enrolled in December 2007.

The study was terminated based on the outcome of the planned first interim analysis, which was performed as defined in the protocol in a subset of patients. It was decided not to continue the trial. No safety concerns were identified.

ELIGIBILITY:
Inclusion Criteria:

* Subject has symptomatic osteoarthritis of the knee diagnosed using clinical and radiographic evidence as well as ACR criteria with symptom duration of at least 6 months.
* Subject requires therapeutic dose of an NSAID, COX-2 NSAID, and/or paracetamol/acetaminophen for osteoarthritis pain of the index knee and has taken that medication at least 5 days per week for the last 4 weeks prior to the screening visit (Visit 1).

Exclusion Criteria:

* Subject is not able to withdraw NSAIDs, COX-2 NSAIDs and/or paracetamol
* Subject is taking analgesic other than NSAIDs COX-2 NSAIDs and/or paracetamol
* Subject is planning to begin or stop treatment with glucosamine and/or chondroitin during the trial

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2007-03; Primary Completion 2007-11 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (26):
- Czechia (2):
  - Kladno
  - Prague
- Germany (5):
  - Bad Hersfeld
  - Berlin
  - Hamburg
  - Leipzig
  - München
- Hungary (6):
  - Debrecen
  - Esztegom
  - Győr
  - Gyula
  - Verseghy
  - Veszprém
- Poland (4):
  - Bialystok
  - Krakow
  - Torun
  - Warsaw
- Romania (4):
  - Brăila
  - Lasi
  - Târgovişte
  - Timișoara
- Stockholm, Sweden
- United Kingdom (4):
  - Morriston
  - Newcastle
  - Oxford
  - Stanmore

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Trial utilized an adaptive 3-stage group sequential design. The Data Monitoring Committee had recommended to stop the trial after the first stage due to lack of efficacy. Results refer to the entire population randomized until discontinuation of study (including overrun).
Pre-assignment Details: Of the 194 enrolled subjects, 149 subjects have been randomized until trial termination. The Participants flow refers to the randomized population. Of the 149 randomized subjects, 148 subjects have been treated and are included in the safety population, 145 have been included in the ITT population (Full Analysis Set).
Groups:
- Lacosamide: Lacosamide (LCM) 400 mg/day
Period: Overall Study
Arm/Group | Lacosamide | Placebo
Started | 73 | 76
Entered Maintenance Phase | 65 | 67
Completed | 57 | 64
Not Completed | 16 | 12
Not completed — Adverse Event | 8 | 5
Not completed — Lack of Efficacy | 5 | 4
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Other | 2 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lacosamide | Placebo | Total
Number analyzed (Participants) | 73 | 76 | 149
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 46 | 86
  >=65 years | 33 | 30 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (8.03) | 62.3 (6.74) | 61.7 (7.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 59 | 111
  Male | 21 | 17 | 38
Region of Enrollment [Number; unit: participants]
  Hungary | 20 | 22 | 42
  Czech Republic | 8 | 10 | 18
  Germany | 27 | 27 | 54
  Poland | 9 | 9 | 18
  Romania | 9 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: Change of the Western Ontario and McMaster Universities (WOMAC) Pain Subscale Score (Visual Analogue Scale Version) From Baseline to the End of the 8 Week Maintenance Period
Description: The Visual Analogue Scale (VAS) version of the WOMAC pain subscale ranges from 0 to 100, high values describe high grade of pain.
Time Frame: Baseline, end of 8 week Maintenance Period
Population: Full Analysis Set (FAS), defined as all randomized subjects that have received at least one dose of trial medication and had at least one post-baseline WOMAC assessment. Last observation carried forward (LOCF) imputation method was applied in case of missing WOMAC assessment.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Lacosamide | Placebo
Number analyzed (Participants) | 71 | 74
Unit on a scale | -24.85 (23.75) | -28.49 (22.27)
Statistical Analysis 1: Comparison: Lacosamide vs Placebo; The ANCOVA analysis includes treatment and pooled site as factors and baseline score as covariate; Test type: Superiority or Other; p = 0.5438, ANCOVA; Mean Difference (Net) = 2.36, 95% CI [-5.30 to 10.02]

2. Secondary Outcome: Change From Baseline to End of 8 Week Maintenance Period in WOMAC Physical Function Subscale Score.
Description: The WOMAC physical function subscale score (Visual Analogue Scale version) ranges from 0 to 100, high values describe high grade of difficulty in performing daily activities.
Time Frame: Baseline, end of 8 week Maintenance Period
Population: Full Analysis Set (FAS), defined as all randomized subjects that have received at least one dose of trial medication and had at least one post-baseline WOMAC assessment. LOCF imputation method was applied in case of missing WOMAC assessment.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Lacosamide | Placebo
Number analyzed (Participants) | 71 | 74
Unit on a scale | -17.09 (21.74) | -23.31 (22.45)
Statistical Analysis 1: Comparison: Lacosamide vs Placebo; The ANCOVA analysis includes treatment and pooled site as factors and baseline score as covariate; Test type: Superiority or Other; p = 0.2022, ANCOVA; Mean Difference (Net) = 4.83, 95% CI [-2.62 to 12.28]

3. Secondary Outcome: Change From Baseline to End of 8 Week Maintenance Period in WOMAC Stiffness Subscale Score.
Description: The WOMAC stiffness subscale score (Visual Analogue Scale version) ranges from 0 to 100, high values describe high grade of stiffness.
Time Frame: Baseline, end of 8 week Maintenance Period
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Lacosamide | Placebo
Number analyzed (Participants) | 71 | 74
Unit on a scale | -18.92 (26.11) | -23.43 (24.00)
Statistical Analysis 1: Comparison: Lacosamide vs Placebo; The ANCOVA analysis includes treatment and pooled site as factors and baseline score as covariate; Test type: Superiority or Other; p = 0.6650, ANCOVA; Mean Difference (Net) = 1.79, 95% CI [-6.36 to 9.93]

4. Secondary Outcome: Change From Baseline to End of 8 Week Maintenance Period in Total WOMAC Score.
Description: The WOMAC total score is the sum of the normalized subscale scores for pain, stiffness, and physical function and ranges from 0 to 300, high values describe high grade of impact.
Time Frame: Baseline, end of 8 week Maintenance Period
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Lacosamide | Placebo
Number analyzed (Participants) | 71 | 74
Unit on a scale | -60.85 (66.85) | -75.24 (65.61)
Statistical Analysis 1: Comparison: Lacosamide vs Placebo; The ANCOVA analysis includes treatment and pooled site as factors and baseline score as covariate; Test type: Superiority or Other; p = 0.3445, ANCOVA; Mean Difference (Net) = 10.74, 95% CI [-11.65 to 33.13]

5. Secondary Outcome: Patient's Global Impression of Change From Baseline at the End of 8 Week Maintenance Period.
Description: Patient's global impression of change from baseline is a score that ranges from 'very much worse' to 'very much improved'.
Time Frame: at the end of 8 week Maintenance Period
Population: Full Analysis Set (FAS), defined as all randomized subjects that have received at least one dose of trial medication and had at least one post-baseline WOMAC assessment. Only subjects with non-missing measurements of Patient's global impression of change from baseline were included.
Measure: Number; unit: Participants
Arm/Group | Lacosamide | Placebo
Number analyzed (Participants) | 68 | 72
Participants
  Very much worse | 4 | 1
  Much worse | 1 | 5
  Worse | 10 | 10
  No change | 18 | 10
  Mildly improved | 12 | 30
  Much improved | 15 | 13
  Very much improved | 8 | 3
  Much + very much improved | 23 | 16
  Much + very much + mildly improved | 35 | 46

6. Secondary Outcome: Response at the End of 8 Week Maintenance Period Versus Baseline Based on the (Slightly Modified)Criteria of the Osteoarthritis Research Society International (OARSI) and the Outcome Measures in Rheumatology Initiative (OMERACT).
Description: Improvement = reduction of >= 20% and >= 10 mm in both WOMAC pain and physical function subscale. Those who met the criteria in either of the subscales had improved if response to Patient's Global Impression of change from baseline was at least 'mildly improved'. High improvement = reduction of >= 50% and >= 20 mm in either of the subscales. Response = either high improvement or improvement.
Time Frame: Baseline, end of 8 week Maintenance Period
Population: Full Analysis Set (FAS), defined as all randomized subjects that have received at least one dose of trial medication and had at least one post-baseline WOMAC assessment. Dropouts due to lack of efficay were defined as non-responders. For dropouts due to any other reason LOCF was applied to the underlying WOMAC subscale scores.
Measure: Number; unit: participants
Arm/Group | Lacosamide | Placebo
Number analyzed (Participants) | 71 | 74
participants
  High improvement | 33 | 32
  Improvement | 38 | 52
  Response | 38 | 52
Statistical Analysis 1: Comparison: Lacosamide vs Placebo; Analysis of 'response' based on a likelihood ratio test with treatment and pooled site as factors; Test type: Superiority or Other; p = 0.0418, Likelihood ratio test; Odds Ratio (OR) = 0.488, 95% CI [0.245 to 0.974]

7. Secondary Outcome: Amount of Rescue Medication Use During 8 Week Maintenance Period.
Description: Use of rescue medication is expressed in number of tablets equivalent to 500 mg Paracetamol per day.
Time Frame: during 8 week Maintenance Period
Population: Full Analysis Set (FAS), defined as all randomized subjects that have received at least one dose of trial medication and had at least one post-baseline WOMAC assessment. Only subjects who entered the Maintenance Phase were included.
Measure: Mean (Standard Deviation); unit: tablets/day
Arm/Group | Lacosamide | Placebo
Number analyzed (Participants) | 65 | 67
tablets/day | 0.48 (0.62) | 0.70 (0.79)

8. Secondary Outcome: Change From Baseline to End of 8 Week Maintenance Period in Perception of Pain Interference With Subject's Sleep.
Description: Pain interference with sleep refers to patient's last evening prior to the visit and was assessed using a 100mm visual analog scale (VAS). The VAS ranges from 0 (did not interfere) to 100 (completely interfered).
Time Frame: Baseline, end of 8 week Maintenance Period
Population: Full Analysis Set (FAS), defined as all randomized subjects that have received at least one dose of trial medication and had at least one post-baseline WOMAC assessment. Only subjects with non-missing values were included.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Lacosamide | Placebo
Number analyzed (Participants) | 57 | 64
Unit on a scale | -19.8 (26.55) | -21.6 (26.76)

9. Secondary Outcome: Change From Baseline to End of 8 Week Maintenance Period in Profile of Mood States (Total Mood Disturbance Score).
Description: Total Mood Disturbance score sums up over the domain scores regarding Tension-anxiety, Depression-ejection, Anger-hostility, Vigor-activity (was subtracted), Fatigue-inertia, Confusion-bewilderment. Domain scores were derived as sum of the respective items and range from 0 to 20. With exception of Vigor-activity high values describe bad mood.
Time Frame: Baseline, end of 8 week Maintenance Period
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Lacosamide | Placebo
Number analyzed (Participants) | 69 | 73
Unit on a scale | 0.9 (17.99) | -4.5 (14.25)

ADVERSE EVENTS:
Arm/Group | Lacosamide | Placebo
Serious Adverse Events (participants affected / at risk) | 4/72 | 2/76
Other Adverse Events (participants affected / at risk) | 16/72 | 13/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lacosamide (N=72) | Placebo (N=76)
Angina pectoris (Cardiac disorders) | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 1 | 0
Liver disorder (Hepatobiliary disorders) | 1 | 0
Shock hypoglycaemic (Metabolism and nutrition disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lacosamide (N=72) | Placebo (N=76)
Vertigo (Ear and labyrinth disorders) | 8 | 1
Fatigue (General disorders) | 4 | 2
Nasopharyngitis (Infections and infestations) | 3 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 4
Headache (Nervous system disorders) | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 days but <= 180 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.